CLINICAL TRIAL: NCT05365737
Title: Substantivity of Mouthrinse Formulations Containing Cetylpyridinium Chloride and O-cymen-5-Ol Compared to Placebo on Salivary Microbiota
Brief Title: Substantivity of Oral Rinses: Comparative Study
Acronym: SORCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Miguel Viñas, Full professor Microbiology, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 33/2021
Record Dates: First submitted 2022-02-23; First posted 2022-05-09 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Prevention & Control
Keywords: Mouth rinses; substanticity; oral infections; salivary microbiota
MeSH Terms: interventions — Mouthwashes

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, crossover study of the in situ antibacterial efficacy of o-Cymen-5-ol plus CPC, o-Cymen-5-ol and CPC on salivary microbiota.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo oral rinse (Placebo Comparator): Placebo comparator Volume Time Active molecule 15 mL 1 min No
  Interventions: Other: Oral rinse; Other: Saliva harvest
- CPC oral rinse (Active Comparator): Volume Time Active molecule 15 mL 1 min CPC containing oral rinse
  Interventions: Other: Oral rinse; Other: Saliva harvest
- Cymenol oral rinse (Active Comparator): Volume Time Active molecule 15 mL 1 min Cymenol containing oral rinse
  Interventions: Other: Oral rinse; Other: Saliva harvest
- CPC + Cymenol oral rinse (Active Comparator): Volume Time Active molecule 15 mL 1 min CPC+cymenol containing oral rinse
  Interventions: Other: Oral rinse; Other: Saliva harvest

INTERVENTIONS:
Other: Oral rinse — Participants use mouthwasher for a given time.
Other: Saliva harvest — Non-stimulated saliva harvesting

SUMMARY:
A desirable quality of mouthrinses is substantivity an intrinsic feature of some molecules. Substantivity requires the adsorption of the agent on the oral surfaces and subsequently antimicrobial activity bacteriostatic along following hours. This work aims to quantitatively determine the substantivity of (i) a single o-Cymen-5-ol plus CPC oral rinse, (ii) a, CPC oral rinse and (iii) a o-Cymen-5-ol mouthwash on the salivary microbiota up to 4 h after their application.

DETAILED DESCRIPTION:
One of the desirable qualities of mouthrinses is substantivity, which is defined as the persistence capacity of its antimicrobial action over time in the mouth. This is an intrinsic feature of some molecules.

Such substantivity seems to require the adsorption of the agent on the buccal surfaces and subsequently exert a certain antimicrobial activity that seems to be mostly bacteriostatic.

Substantivity is the result of multiple factors controlling or altering adhesion, life period of antimicrobial capabilities, synergisms, antagonisms, and others. In order to improve substantivity and therefore increase antimicrobial effectiveness of CPC, o-Cymen-5-ol has recently been proposed to become incorporated to oral rinses. The aim of this work is to quantitatively determine the substantivity of (i) a single o-Cymen-5-ol plus CPC oral rinse, (ii) a, CPC oral rinse and (iii) a o-Cymen-5-ol mouthwash on the salivary microbiota up to 4 h after their application.

ELIGIBILITY:
Inclusion criteria:

1. adult age (>18 y/o)
2. good oral helath status
3. minimum 24 evaluable teeth
4. periodontal pockets ≤3 mm
5. absence of caries & periodontal haemorrage

Exclusion Criteria:

1. smokers
2. prosthesis or orthodontic devices
3. Sjögren syndrome
4. Antibiotic treatment in the last three months
5. Systemic disease with alteration in the production and/or composition of the saliva

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Preliminary experiments | one month
  Measure of surviving bacteria by fluorimetry and confocal microscopy (Live & dead)

SECONDARY OUTCOMES:
Substantivity of mouthrinse formulations containing Cetylpyridinium Chloride and O-cymen-5-Ol (single and combined) compared to Placebo on salivary microbiota | up to three months
  Measure of surviving bacteria by fluorimetry and confocal microscopy (Live & dead) rinses plus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Viñas, PhD, Study Chair — University of Barcelona-Spain-
Locations (1):
- University of Barcelona. Campus Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aguilera FR, Vinas M, Sierra JM, Vinuesa T, R Fernandez de Henestrosa A, Furmanczyk M, Trullas C, Jourdan E, Lopez-Lopez J, Jorba M. Substantivity of mouth-rinse formulations containing cetylpyridinium chloride and O-cymen-5-ol: a randomized-crossover trial. BMC Oral Health. 2022 Dec 27;22(1):646. doi: 10.1186/s12903-022-02688-z. PMID 36575444